CLINICAL TRIAL: NCT03546335
Title: Zirconium-89 Certolizumab PET Imaging in Patients With Rheumatoid Arthritis
Brief Title: Zr-89 Cimzia PET Imaging Rheumatoid Arthritis
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: Lapse in study funding.
Sponsor: Robert Flavell, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Robert Flavell, MD, PhD, Assistant Professor in Residence, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 17-23566
Record Dates: First submitted 2018-04-30; First posted 2018-06-06 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Intervention Model Description: The first 2 patients will receive 1 mCi of 89Zr-DFO-CZP. Subsequent groups of two patients will receive 0.5 mCi decrease or increase dose (up to 2 mCi) to determine the acceptable optimal imaging dose.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 1 mCi injection of 89Zr-DFO-CZP (Experimental): The first 2 patients will receive 1 mCi of 89Zr-DFO-CZP.
  Interventions: Drug: 89Zr-DFO-CZP
- 0.5 mCi injection of 89Zr-DFO-CZP (Experimental): Subsequent groups of two patients will receive 0.5 mCi decrease or increase dose (up to 2 mCi) to determine the acceptable optimal imaging dose.
  Interventions: Drug: 89Zr-DFO-CZP
- 1.5 mCi injection of 89Zr-DFO-CZP (Experimental): Subsequent groups of two patients will receive 0.5 mCi decrease or increase dose (up to 2 mCi) to determine the acceptable optimal imaging dose.
  Interventions: Drug: 89Zr-DFO-CZP
- 2 mCi injection of 89Zr-DFO-CZP (Experimental): Subsequent groups of two patients will receive 0.5 mCi decrease or increase dose (up to 2 mCi) to determine the acceptable optimal imaging dose.
  Interventions: Drug: 89Zr-DFO-CZP

INTERVENTIONS:
Drug: 89Zr-DFO-CZP — 89Zr-DFO-Certolizumab pegol (89Zr-DFO-CZP) is a radiopharmaceutical imaging agent that will be produced under Current Good Manufacturing Practice (CGMP) regulations in the Department of Radiology and Biomedical Imaging Radiopharmaceutical Facility at University of California, San Francisco (UCSF).
  Other Names: 89Zr-Cimzia

SUMMARY:
This is a single center exploratory imaging study investigating the initial application of zirconium-89 Deferoxamine B Certolizumab pegol (89Zr-DFO-CZP) PET in patients with rheumatoid arthritis. Patients with active symptoms of RA or signs on physical exam will be invited to participate for PET imaging.

DETAILED DESCRIPTION:
This is a single center exploratory imaging study investigating the initial application of 89Zr-DFO-CZP PET in patients with rheumatoid arthritis. Patients with active symptoms of rheumatoid arthritis (RA) or signs on physical exam will be invited to participate for PET imaging. Study 1 is a dose finding study that will involve a single 89Zr-DFO-CZP PET scan acquired ~24 hours following a single administration of the radiopharmaceutical. The first 2 patients will receive 1 millicurie (mCi) of 89Zr-DFO-CZP. Subsequent groups of two patients will receive 0.5 mCi decrease or increase dose (up to 2 mCi) to determine the acceptable optimal imaging dose. After receiving the dose, participants will undergo 4 serial whole body PET scans between 2 hours and 120 hours after dose administration. Several blood samples will also be collected over this time period, for dosimetry analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years old.
2. Ability to read and understand written informed consent document.
3. Patients with clinical diagnosis of rheumatoid arthritis.

Exclusion Criteria:

1. For patients planning to be imaged on PET (positron emission tomography) / MRI (magnetic resonance imaging) (PET/MR) scanner, exclusion criteria will include any contra-indication to MRI, including permanent pacemaker, implantable metallic device/ prosthetic, aneurysm clip, non-removable piercing, or severe claustrophobia.
2. Any medical condition that would compromise the imaging acquisition, in the opinion of the investigator.
3. Patients who have had a study involving radiation within one year of enrolling in this study.
4. Patients who are pregnant (female patients of childbearing age will be tested prior to injection of imaging agent - positive test will exclude from participating in the study).
5. Patients who are breastfeeding.
6. Patients who cannot confirm that they will use reliable contraceptive methods for 90 days.
7. Patients treated with TNF-alpha inhibitor therapy.
8. Females of child-bearing age (<50 years old), until data from the dose-finding study has been reviewed by the UCSF Radiation Safety Committee and explicit written permission has been provided by the UCSF Radiation Safety Committee to open the window of potential female participants to ages 18 years and older.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Uptake of 89Zr-DFO-CZP taken up in symptomatic versus asymptomatic joints of patients with rheumatoid arthritis (RA). | 2 years
  Investigators will be evaluating whether 89Zr-DFO-CZP is taken up in symptomatic versus asymptomatic joints of patients with rheumatoid arthritis (RA).

SECONDARY OUTCOMES:
Uptake of 89Zr-DFO-CZP in symptomatic joints of patients with rheumatoid arthritis after administration of a Tumour Necrosis Factor alpha (TNF-alpha) inhibitor therapeutic. | 2 years
  Investigators will be evaluating the uptake of 89Zr-DFO-CZP in symptomatic joints of patients with rheumatoid arthritis after administration of a TNF-alpha inhibitor therapeutic.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Flavell, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No